CLINICAL TRIAL: NCT00085423
Title: High Dose Interleukin-2 (IL-2) Therapy In "Lymphodepleted Primed" Patients With Metastatic Melanoma
Brief Title: Cyclophosphamide, Fludarabine, and High-Dose Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000370788; P30CA023108 (NIH); DMS-0320 (Other: Dartmouth-Hitchcock); DMS-16531 (Other: Dartmouth-Hitchcock); NCT00225771 (obsolete NCT alias)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Interleukin-2; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IL-2, CTX, fludarabine, GM-CSF (Experimental): Aldesleukin (IL-2), cyclophosphamide, fludarabine phosphate, sargramostim
  Interventions: Biological: aldesleukin; Biological: sargramostim; Drug: cyclophosphamide; Drug: fludarabine phosphate

INTERVENTIONS:
Biological: aldesleukin — ‡Interleukin-2 (aldesleukin) IV (600,000 U/kg; Chiron, Emeryville, CA): two 5-day courses on days 8 and 22. Interleukin-2 was given over 15 minutes every 8 hours. Goal is 14 doses/5-day course
  Other Names: Aldesleukin; IL-2; HD IL-2; Interleukin-2
Biological: sargramostim — GM-CSF was given subcutaneously daily from day 8 until absolute granulocyte count exceeds 5,000 cells/mL for 2 consecutive days.
  Other Names: GM-CSF; granulocyte-macrophage colony-stimulating factor
Drug: cyclophosphamide — Cyclophosphamide (60 mg/kg/d; Baxter, Deerfield, IL) intravenously (IV) for 2 days with sodium 2- mercaptoethanesulfonate (Mesna; Sicor, Irvine, CA) at 20% of cyclophosphamide dose IV 15 minutes before and 40% of the cyclophosphamide dose orally at 2 and 6 hours after the initiation of chemotherapy.
  Other Names: cyclophosphamide,Cytoxan
Drug: fludarabine phosphate — Fludarabine IV (25 mg/M2/day)-five daily doses from Day 3
  Other Names: Fludara

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide and fludarabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: This phase II trial is studying how well giving cyclophosphamide and fludarabine together with high-dose interleukin-2 works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in lymphodepleted patients with metastatic melanoma treated with cyclophosphamide, fludarabine, and high-dose interleukin-2.
* Determine the feasibility of this regimen in these patients.

Secondary

* Determine the quality and quantity of lymphocyte recovery in these patients during and after treatment with this regimen.
* Determine time to disease progression and survival in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive lymphodepleting therapy comprising cyclophosphamide IV over 1 hour on days 1 and 2 and fludarabine IV over 30 minutes on days 3-7. Patients then receive high-dose interleukin-2 IV every 8 hours (14 doses) on days 8-12 and 22-26. Patients also receive sargramostim (GM-CSF) subcutaneously beginning on day 8 and continuing until blood counts recover. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-33 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma
* Metastatic disease
* Measurable disease
* No history of brain metastases
* Over 18
* Karnofsky 60-100%
* Life expectancy At least 12 weeks
* Hematopoietic
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.5 g/dL
* aspartate aminotransferase ≤ 2 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin ≤ 2 times ULN (except for patients with Gilbert's syndrome)
* Hepatitis B and C negative
* Creatinine ≤ 2.0 times ULN
* Creatinine clearance ≥ 50 mL/min
* Cardiovascular
* Ejection fraction ≥ 50%
* No evidence of congestive heart failure
* No symptoms of coronary artery disease
* No serious cardiac arrhythmias
* No myocardial infarction within the past 6 months
* Cardiac stress test negative or of low probability for patients > 40 years of age OR who have had prior myocardial infarction > 6 months ago
* Pulmonary Forced expiratory volume 1 ≥ 2.0 liters OR at least 75% of predicted for height and age
* Diffusing capacity of lung for carbon monoxide ≥ 60%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

Exclusion Criteria:

* No uncontrolled diabetes
* No history of autoimmune disease
* No active infection
* No other concurrent significant illness that would preclude study participation
* No other malignancy within the past 5 years except nonmelanoma skin cancer or non-invasive cancer (e.g., carcinoma in situ of the cervix, superficial bladder cancer without local recurrence, or carcinoma in situ of the breast)
* At least 4 weeks since prior immunotherapy and recovered
* No other concurrent anticancer biologic agents
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent chemotherapy
* At least 4 weeks since prior steroid therapy
* No concurrent corticosteroids
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy
* At least 4 weeks since prior surgery and recovered
* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-02; Primary Completion 2008-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc S. Ernstoff, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Result] Gunturu KS, Meehan KR, Mackenzie TA, Crocenzi TS, McDermott D, Usherwood EJ, Margolin KA, Crosby NA, Atkins MB, Turk MJ, Ahonen C, Fuse S, Clark JI, Fisher JL, Noelle RJ, Ernstoff MS. Cytokine working group study of lymphodepleting chemotherapy, interleukin-2, and granulocyte-macrophage colony-stimulating factor in patients with metastatic melanoma: clinical outcomes and peripheral-blood cell recovery. J Clin Oncol. 2010 Mar 1;28(7):1196-202. doi: 10.1200/JCO.2009.24.8153. Epub 2010 Feb 1. PMID 20124177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment was open from February 2004 to December 2008.
Groups:
- Lymphodepleting Chemotherapy + High Dose Interleukin-2: Lymphodepleting chemotherapy + high dose interleukin-2:
  Intravenous cyclophosphamide (60 mg/kg, days 1 and 2) and fludarabine (25 mg/m(2), day 3 through 7) followed by two 5-day courses of intravenous high-dose bolus IL-2 (600,000 U/kg; days 8 through 12 and 21 through 25). Granulocyte-macrophage colony-stimulating factor, GM-CSF, (250 microg/m(2)/d beginning day 8) was given until granulocyte recovery.
Period: Overall Study
Arm/Group | Lymphodepleting Chemotherapy + High Dose Interleukin-2
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — screen failure | 1

BASELINE CHARACTERISTICS:
Groups:
- Lymphodepleting Chemotherapy + High Dose IL-2: intravenous cyclophosphamide (60 mg/kg, days 1 and 2) and fludarabine (25 mg/m(2), day 3 through 7) followed by two 5-day courses of intravenous high-dose bolus IL-2 (600,000 U/kg; days 8 through 12 and 21 through 25). GM-CSF (250 microg/m(2)/d beginning day 8) was given until granulocyte recovery.
Arm/Group | Lymphodepleting Chemotherapy + High Dose IL-2
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of partiCIPANTS WITH OBJECTIVE RESPONSE AS MEASURED BY RECIST
Description: Objective response as measured by radiological and physical examination using RECIST criteria.
Time Frame: Response at 12 weeks
Population: Response was determined by physical examination and radiologic testing. Percent of the total number of patients treated was calculated.
Measure: Number; unit: participants
Groups:
- Group 1: all patients are treated with lymphodepleting chemotherapy and highdose IL-2 and GM-CSF.
Arm/Group | Group 1
Number analyzed (Participants) | 18
participants | 3

2. Secondary Outcome: Number of Participants With Lymphocyte Recovery as Measured by Blood Count
Description: Lymphocyte recovery to a greater than 1000 cells/mcL was determined by differential peripheral blood cell counts on sequential days as noted in time frame.
Time Frame: on days 1-15, weekly for 2 weeks, and then every 2-3 months
Population: each patient's differential blood counts were used to determine the time of recovery to the lower limit of normal lymphocytes in the peripheral blood.
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 18
participants | 18 [1000 to 4000]

3. Secondary Outcome: Time to Progression as Measured by RECIST
Description: Clinical outcome used the National Cancer Institute's Response Evaluation Criteria in Solid Tumors (RECIST)1.0.
Time Frame: From date of randomization until the first date of documented progression or date of death from any cause, which ever came first, assessed up till 100 months
Measure: Mean (95% Confidence Interval); unit: years
Arm/Group | Group 1
Number analyzed (Participants) | 18
years | .3 [.2 to .4]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 8/18
Other Adverse Events (participants affected / at risk) | 4/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=18)
anemia (Blood and lymphatic system disorders) | 8 (18) — 8 patients required blood transfusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=18)
thrombocytopenia (Blood and lymphatic system disorders) | 4 (18) — 4 patients required platelet transfusion

LIMITATIONS AND CAVEATS:
This was the first stage of a two-stage phase II study and continuation to next stage required 4 of 18 particpant having an objective response. Only 3 objective responses were noted and the study was terminated at stage 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No